CLINICAL TRIAL: NCT00886106
Title: The Effect of High-dose Remifentanil on Established Capsaicin-induced Hyperalgesia in Human Volunteers
Acronym: RemiAnes 1
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Professor Burkhard Gustorff, Medical University of Vienna, Dept. Anaesthesia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: RemiAnes 1
Record Dates: First submitted 2009-04-21; First posted 2009-04-22 (Estimated); Last update posted 2009-11-18 (Estimated); Status verified 2009-11

CONDITIONS: Hyperalgesia
Keywords: Capsaicin; Remifentanil; Hyperalgesia
MeSH Terms: conditions — Hyperalgesia | interventions — Remifentanil; Midazolam

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Remifentanil
  Interventions: Drug: Remifentanil
- 2 (Active Comparator): Midazolam
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Remifentanil — Remifentanil (Ultiva®; Glaxo-Smith-Kline; Vienna, Austria) will be applied intravenously during 60 minutes through a dedicated infusion pump (TCI Alaris PK Syringe Pump, Cardinal Health, Baesweiler, Germany), with a Target Controlled Infusion (following the integrated software algorithm by Minto), reaching the initial 18ng/ml plasma concentration in 180 seconds. This corresponds to circa 0.7 µg kg-1 min-1
  Arms: 1
Drug: Midazolam — Midazolam (Dormicum®; Roche; Vienna, Austria) will be applied intravenously as active placebo at a dose of 15 µg kg-1 min-1 over 5 minutes to mimic typical central nervous side effects of remifentanil
  Arms: 2

SUMMARY:
Treatment of chronic pain is a major clinical challenge since chronic pain is frequent and leads to deterioration of quality of life. An injury or wound can lead to long term changes in the nervous system that make the skin more sensitive at and near the injury; this is termed hyperalgesia and occurs through long term depotentiation (LTP), i.e., a change in the synaptic interaction between neurons.

Opioids are the gold standard for the symptomatic therapy of moderate to severe pain. Now, in animal studies the investigators have discovered previously unrecognized effects of opioids.

Intradermal injection of capsaicin (injection of pepper extract into the skin) is an established pain model in humans. The investigators want to test the influence of remifentanil, an ultra-short acting opioid, on hyperalgesia observed after intradermal capsaicin in human volunteers in a double blind cross-over prospective active placebo controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Men or women, aged between 19 and 40 years
* Body mass index between 15th and 85th percentile
* Normal findings in the medical history and physical examination
* Drug free for 1 week prior to the study day

Exclusion Criteria:

* Regular use of medication especially analgesics
* Abuse of alcoholic beverages, drug abuse
* History of asthma
* Participation in a clinical trial in the 2 weeks preceding the study
* Symptoms of a clinically relevant illness in the 2 weeks before the first study day
* Resting systolic blood pressure > 135 mmHg or diastolic blood pressure > 85 mmHg
* Acute skin diseases like sunburn on the relevant areas or skin lesions
* Pregnancy or breast feeding
* Regular consumption of very spicy (capsaicin containing) food
* Allergy against any medication used in the study protocol

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2009-06; Primary Completion 2009-12 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Area of pin prick hyperalgesia | 0-6 hours

SECONDARY OUTCOMES:
Pain immediately after injection | 0-15 min
Stimulus-response (SR) function to a set of modified rigid von Frey filaments (8-512 mN) | 0-6 hours
Heat pain threshold within the area of mechanical hyperalgesia | 0-6 hours
Mechanical pain threshold within the area of pin prick hyperalgesia, area of dynamic allodynia to brush | 0-6 hours
Adverse effects | 30 and 59 min after infusion of study medication

CONTACTS AND LOCATIONS:
Overall Officials: Burkhard Gustorff, MD, Study Chair — Medical University of Vienna
Locations (1):
- Department of Anaesthesia, Medical University of Vienna, Vienna, Vienna, Austria